CLINICAL TRIAL: NCT05883033
Title: Comparative Study Between Vacuum Assisted Closure (VAC) and Conventional Dressing in the Healing Process of Necrotizing Fasciitis After Surgical Debridement.. Clinical and Laboratory Study.
Brief Title: VAC and Conventional Dressing in the Healing Process of Necrotizing Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mario Youhana Saba, Resident Dr, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Necrotizing fasciitis
Record Dates: First submitted 2023-04-22; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Necrotizing Fascitis
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum Assisted Closure device (Experimental): Vacuum Assisted Closure device for healing enhancement
  Interventions: Device: VAC
- Conventional dressing (Experimental): Unprocessed Honey, malysia glycerine and betadine ointment
  Interventions: Device: VAC

INTERVENTIONS:
Device: VAC — Vacuum Assisted Closure device

SUMMARY:
Find out the best management of Necrotizing Fasciitis after surgical debridement

DETAILED DESCRIPTION:
Necrotizing fasciitis is a life-threatening condition that can occur as a result of trauma or foreign bodies in surgical wounds as well as idiopathically. Necrotizing fasciitis is characterized by a progressive infection in fascial planes with necrosis of the subcutaneous tissue. Necrotizing fasciitis affects the extremities more frequently than central areas. Risk factors for necrotizing fasciitis include diabetes mellitus, trauma wound infections, decubitus ulcers, alcoholism, carcinoma, peripheral vascular disease, smoking, and intravenous drug abuse. A varieties of micro-organisms, including gram-positive group A streptococcus, haemolytic streptococci, and staphylococcus aureus; gram-negative Enterobacteriaceae, Escherichia coli, Klebsiella spp., and Proteus spp.; anaerobes including Peptostreptococcus, Clostridium, and Pacteroides; and fungi such as Candida and acid-fast bacteria have all been implicated in the pathogenesis of Necrotizing fasciitis.

Necrotizing fasciitis is a surgical emergency for detoxification by debridement with good antibiotic coverage. It has mortality rate reaching 20-30% , this mortality rate is high and requires prompt diagnosis, antibiotic treatment and extensive necrosectomy up to intensive care units admission in some cases, the aim of our prospective analysis is to assess with a hypothesis-generating and exploratory purpose the possible role of VAC versus ordinary dressings in the wound therapy of Necrotizing Fasciitis in terms of expected time for wound closure and survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patients such as; diabetic, HIV and leukaemia.

And other chronic debilitating diseases.

Exclusion Criteria:

* Necrotizing Fasciitis of Head and neck and upper limbs.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Hospital staying length | Baseline
  the difference in hospital stay length between patients with necrotizing fasciitis who received conventional management versus those treated with vacuum-assisted closure. A systematic review showed a significant difference between the two methods

SECONDARY OUTCOMES:
Required other stages of debridement | Baseline
  Comparison in the other stages of debridement required in both methods
Expected closure of the wound by secondary intention | Baseline
  The difference in expected time required for closure of the wound by secondary intention between patients with necrotizing fasciitis who received conventional management versus those treated with vacuum-assisted closure.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang R, Zhang Y, Hou L, Yan C. Vacuum-assisted closure versus conventional dressing in necrotizing fasciitis: a systematic review and meta-analysis. J Orthop Surg Res. 2023 Feb 4;18(1):85. doi: 10.1186/s13018-023-03561-7. PMID 36737764